CLINICAL TRIAL: NCT00922142
Title: Cesarean Postoperative Pain Satisfaction With Intravenous Patient-Controlled Analgesia Intravenous, Oral, or Epidural Method
Brief Title: Cesarean Postoperative Pain Satisfaction
Status: Completed | Type: Observational
Sponsor: Saint Elizabeth Regional Medical Center (Other)
Responsible Party: Debbie Cahmber/Director Perinatal Nursing, Saint Elizabeth Regional Medical Center
Other Study IDs: 608-028
Record Dates: First submitted 2009-06-16; First posted 2009-06-17 (Estimated); Last update posted 2011-07-20 (Estimated); Status verified 2011-07

CONDITIONS: Cesarean

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — no biospecimens to be retained
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Hypothesis:

There is no significant difference in Cesarean patients' perceptions of overall pain management satisfaction between methods used for postoperative pain management.

DETAILED DESCRIPTION:
There is a significant difference between Cesarean patients' perceptions of advantages and disadvantages of three postoperative pain management methods identified by obstetrical patients.

Participants will be introduced to study by anesthesia personnel in labor and delivery. The subject will be informed of the desire for their input on their perceived satisfaction with their chosen method for post-operative pain management and will be asked to participate in an anonymous survey by their second day after surgery. They will be informed that this is voluntary. Method of post-operative medication administration will be determined by attending physician to be either: epidural, IVPCA, or oral medication. Methods will be initiated in recovery room or the operative suite.

Subjects will be identified on a postpartum admission log and a screening log will be created for study purposes.

Informed Consents will be obtained. The screening log entries will be numbered corresponding to a numbered survey. The screening log will contain demographic and other patient identifiers including age, ethnicity, parity, presence of labor prior to cesarean, admission status of baby, cost associated with method and presence of rescue drugs and costs of rescue drugs and method services. Refusal information, exclusion criteria, and time/date of survey completion will also be recorded. This log will be maintained under lock and key.

ELIGIBILITY:
Inclusion Criteria:

* English speaking post-operative cesarean patients

Exclusion Criteria:

* Cesarean patients with know fetal demise
* General/Local Anesthetic Method for Cesarean

Ages: 14 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: post-operative cesarean patients
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2009-06; Primary Completion 2009-08 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deb Chambers, RN, Principal Investigator — Saint Elizabeth Regional Medical Center
Locations (1):
- Saint Elizabeth Regional Medical Center, Lincoln, Nebraska, United States